CLINICAL TRIAL: NCT03633812
Title: The Effect of Preoperative Beta Blocker Use on Intraoperative Hemodynamics and Postoperative Renal Function in End-stage Liver Disease Patients Undergoing Liver Transplantation
Brief Title: Effect of Preoperative Beta Blocker Use Postoperative Renal Function in the Patients Undergoing Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jun-Gol Song, Professor, Asan Medical Center
Other Study IDs: 2016-1159
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: End Stage Liver Disease; Acute Kidney Injury
Keywords: End Stage Liver Disease; Acute Kidney Injury; Beta blocker
MeSH Terms: conditions — End Stage Liver Disease; Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beta blocker group: ESLD recipients who had beta blocker during more than 1 month before the liver transplantation
  Interventions: Other: Observational study, Beta blocker medication history
- Non-Beta blocker group: ESLD recipients who had not taken beta blocker more than 3 month before the liver transplantation

INTERVENTIONS:
Other: Observational study, Beta blocker medication history — Observational study, Beta blocker medication history
  Groups: Beta blocker group

SUMMARY:
This is prospective cohort study of patients classified by the premedication history of beta-blocker. The investigators aim to evaluate the hemodynamic effect of beta blocker through Swan-Ganz catheter monitoring and arterial pressure waveform analysis during surgery. The investigators also plan to observe the long-term effects of beta blocker on acute renal failure, allograft failure and mortality.

DETAILED DESCRIPTION:
Since beta blockers have been shown to reduce portal venous pressure in 1980, the nonselective beta blocker (NSBB) has been widely used for the last 25 years as the primary treatment for portal hypertension. NSBB, such as propranolol and nadolol, has been shown to reduce cardiac output through β1 -receptor block and to constrict visceral vessels via β2-receptor block, thereby lowering portal venous pressure in patients with chronic liver disease. NSBB contributed to reducing complications such as esophageal variceal bleeding, ascites, hepatic encephalopathy, and improving survival in patients with cirrhosis. In addition, the use of NSBB in patients with ascites has been demonstrated to reduce the digestion time of intestinal food and reduce bacterial migration into the abdominal cavity and bloodstream.

On the other hand, recent studies have shown that NSBB use in the patients with advanced cirrhosis (accompanied by refractory ascites, spontaneous peritonitis, severe alcoholic hepatitis) may increase circulatory failure, acute renal failure, and mortality. When the cardiac index was less than 1.5 L / min / m² or the mean blood pressure was less than 80 mmHg in advanced cirrhosis with ascites, 1-year survival rate was found to be about 30% lower than the control. The use of beta blockers is argued to be avoided in the cirrhotic patients with refractory ascites because the mortality rate of these patients is associated with the use of beta blockers. These studies have been questioned in terms of reliability of the setting of treatment and control groups and correction of disturbance variables.

The window hypothesis has received attention for the risk-benefit of NSBB. This means that the beta blocker may be beneficial or harmful to the cirrhotic patients depending on the stage of disease progression. In conclusion, the use of beta-blockers in patients with early cirrhosis without moderate to large varix has no effect on prevention of esophageal varices, but is associated with depression, tiredness, sexual dysfunction, decreased cardiac output, increased risk of heart failure, symptomatic bradycardia, increased airway resistance, and bronchospasm. As the cirrhosis progresses, many changes occur in the cardiovascular system. The sympathetic nervous system and resin-angiotensin-aldosterone axis are up-regulated to compensate for the lack of effective blood volume due to peripheral vascular relaxation and hypotension. It is believed that the use of beta-blockers at this time may improve survival by reducing esophageal bleeding and bacterial migration. If the liver cirrhosis progresses more, the use of beta-blockers may compromise cardiac output, blood pressure, perfusion to important organs, thereby increasing the incidence of hepatorenal syndrome and mortality. The use of beta-blockers seems to be beneficial between the point of moderate to large varix generation to the point of advanced cirrhosis with undesired hemodynamic effect (spontaneous ascites, hepatorenal syndrome, spontaneous bacterial peritonitis, sepsis). The research is still ongoing and controversial.

As mentioned earlier, the use of beta blockers in patients with liver disease has been actively studied for the last 10 years, but most studies have been done in patients waiting for liver transplantation. Research is minimal in patients who actually undergo liver transplantation. In addition, studies have shown that beta blockers increase survival in patients waiting for liver transplantation by lowering portal venous pressure through beta 1, 2 -receptor block. But the actual research of preoperative beta blocker on perioperative hemodynamics, postoperative complications, and mortality is still lacking.

This is prospective cohort study of patients classified by the premedication history of beta-blocker. The investigators aim to evaluate the hemodynamic effect of beta blocker through Swan-Ganz catheter monitoring and arterial pressure waveform analysis during surgery. The investigators also plan to observe the long-term effects of beta blocker on acute renal failure, allograft failure and mortality.

ELIGIBILITY:
Inclusion Criteria:

* living donor liver transplantation recipients

Exclusion Criteria:

* previous history of acute kidney injury
* previous liver transplantation history
* Fulminant hepatic failure
* history of TIPS, transjugular intrahepatic porto-systemic shunt

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: living donor liver transplant recipients at Asan Medical Center, Seoul, Korea, Republic of
Sampling Method: Non-Probability Sample
Enrollment: 477 (Estimated)
Dates: Start 2016-10-28 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 1 week
  Creatinine change

SECONDARY OUTCOMES:
Graft failure | 1 year
  Graft failure
Mortality | 1 year
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jun Gol Song, PH.D., Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Asan medical center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krag A, Wiest R, Albillos A, Gluud LL. The window hypothesis: haemodynamic and non-haemodynamic effects of beta-blockers improve survival of patients with cirrhosis during a window in the disease. Gut. 2012 Jul;61(7):967-9. doi: 10.1136/gutjnl-2011-301348. Epub 2012 Jan 10. No abstract available. PMID 22234982
- [Background] Serste T, Melot C, Francoz C, Durand F, Rautou PE, Valla D, Moreau R, Lebrec D. Deleterious effects of beta-blockers on survival in patients with cirrhosis and refractory ascites. Hepatology. 2010 Sep;52(3):1017-22. doi: 10.1002/hep.23775. PMID 20583214
- [Background] Serste T, Francoz C, Durand F, Rautou PE, Melot C, Valla D, Moreau R, Lebrec D. Beta-blockers cause paracentesis-induced circulatory dysfunction in patients with cirrhosis and refractory ascites: a cross-over study. J Hepatol. 2011 Oct;55(4):794-9. doi: 10.1016/j.jhep.2011.01.034. Epub 2011 Feb 24. PMID 21354230